CLINICAL TRIAL: NCT04988243
Title: Multi Center Registry of Transcatheter Aortic Valve Replacement in Northeast China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CCRF Inc., Beijing, China (Industry)
Collaborators: Hangzhou Qiming Medical Instrument Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Yaling Han, M.d., Ph.D., Academlcan/chief physician, CCRF Inc., Beijing, China
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB001
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Severe Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Retrospective subjects were subjects who had completed transcatheter aortic valve replacement at the beginning of the study. Previous data such as demography and treatment of subjects before the start of the study will be realized by reviewing medical records. Follow up data not traceable to medical records and follow-up data after the start of the study, Prospective subjects were those who were undergoing or planned to undergo transcatheter aortic valve replacement at the beginning of the study. Subjects were enrolled from the beginning of the first case to one year later. The demographic, treatment and follow-up data of subjects will be collected through clinical follow-up or telephone follow-up
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective and retrospective study of subjects undergoing aortic valve surgery (Other): This study is a prospective / retrospective, multicenter, and observational study after listing. The researchers can initially determine that they can be enrolled in the study according to the history diagnosis of the subjects. After fully informed, they sign informed consent form. After the evaluation of the researchers, they meet the TAVR selection requirements, and register the subjects in multiple centers at the same time
  Interventions: Other: All aortic valve products on the market

INTERVENTIONS:
Other: All aortic valve products on the market — 1. Subjects with severe aortic valve stenosis
  2. Subjects who plan (or have) to use the transcatheter aortic valve replacement system for percutaneous aortic valve replacement
  3. The patients agreed to join the study, voluntarily signed the informed consent and completed the follow-up;
  4. Be able to contact the subjects or their legal guardians / relatives;
  5. The medical record records the subjects who have died and can't get any contact information of the subjects（ (for dead cases only)
  Sign the informed consent form, then check the inclusion and exclusion criteria, register after meeting the criteria, obtain the registration number, perform aortic valve replacement surgery, follow-up 24 hours, discharge, 30 days, 1 year, 2 years, 3 years, 4 years and 5 years after operation according to the test requirements, and carry out relevant follow-up according to the scheme requirements to collect data

SUMMARY:
The purpose of this study was to observe the safety and effectiveness of transcatheter aortic valve replacement in patients with aortic valve stenosis in a real-world clinical practice environment.

DETAILED DESCRIPTION:
This study is a prospective / retrospective, multicenterstudy after listing. The researchers preliminarily confirmed that they could be enrolled in this study according to the diagnosis of the subjects' medical history. After fully informed, they signed the informed consent, and met the TAVR inclusion requirements (see the inclusion criteria for details). At the same time, they registered the subjects in multiple centers. After the start of the trial, the participants were enrolled in the study, All the subjects who met the inclusion criteria but did not meet the discharge criteria were registered in the central registration system. The patients were followed up for 30 days, 6 months and 12 months, and followed up by telephone for 2, 3, 4 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic valve stenosis, defined as follows:

   1. Symptomatic patients:

      * The mean differential pressure measured by echocardiography ≥ 40mm Hg
      * Or peak aortic ejection ≥ 4.0 m / S
      * Or aortic valve area ≤ 1.0cm ²（ Or AVA index ≤ 0.6 cm2 / m2)
   2. Asymptomatic patients:

      * Severe aortic stenosis and aortic valve area ≤ 1.0cm ²（ 6 cm2 / m2) with aortic ejection peak value ≥ 5.0 M / s or mean pressure difference measured by --echocardiography ≥ 60 mm Hg;
      * Or aortic valve area ≤ 1.0cm ²（ Or AVA index ≤ 0.6 cm2 / m2), combined with aortic ejection peak ≥ 4.0 m / s or average differential pressure measured by echocardiography ≥ 40 mm Hg, combined with limited exercise tolerance test, abnormal blood pressure response or arrhythmia;
      * Or aortic valve area ≤ 1.0cm ²（ Or AVA index ≤ 0.6 cm2 / m2), combined with aortic ejection peak ≥ 4.0 m / s or average differential pressure measured by echocardiography ≥ 40 mm Hg, combined with LVEF < 50%
2. Subjects who plan (or have) to use the transcatheter aortic valve replacement system for percutaneous aortic valve replacement
3. The patients agreed to join the study, voluntarily signed the informed consent and completed the follow-up;
4. Be able to contact the subjects or their legal guardians / relatives;
5. The medical record records the subjects who have died and can't get any contact information of the subjects（ (for dead cases only)

Note: for dead subjects, they must meet 1, 2 and 5 at the same time before they can be included in the group.

Exclusion Criteria:

1. Contraindications to any artificial biological valve implantation;
2. Any known allergies or contraindications;

   * Aspirin or heparin and bivalirudin;
   * Tigrelol and clopidogrel;
   * Nickel titanium alloy;
   * Contrast medium;
3. The patient is currently participating in drug or device research;
4. The patient is pregnant or lactating;
5. Aortic annulus diameter < 17 mm or > 32 mm;
6. The diameter of approach vessel was less than 5.0mm;
7. The investigator believes that the patient is not suitable to participate in this study or complete the follow-up specified in the protocol;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Primary end point: the incidence of all-cause death 12 months after operation | 12 months after aortic valve replacement
  After subjects completed aortic valve replacement surgery, whether prospectively or retrospectively, all-cause mortality at 12 months after operation was collected according to the time node of subjects' enrollment

SECONDARY OUTCOMES:
The compound incidence of death, surgery, severe stroke, life-threatening bleeding, serious vascular complications and acute renal failure (within 30 days after operation); | Within 30 days after aortic valve replacement
  The compound incidence of death, surgery, severe stroke, life-threatening bleeding, serious vascular complications and acute renal failure (within 30 days after operation);
The implantation rate of permanent pacemaker within 30 days; | Within 30 days after aortic valve replacement
  The implantation rate of permanent pacemaker within 30 days;
All stroke (disabled or not disabled) within 12 months and 2, 3, 4 and 5 years | 12 months and within 2, 3, 4 and 5 years
  All stroke (disabled or not disabled) within 12 months and 2, 3, 4 and 5 years;
the incidence of life-threatening bleeding within 12 months and 2, 3, 4 and 5 years; | 12 months and within 2, 3, 4 and 5 years
  the incidence of life-threatening bleeding within 12 months and 2, 3, 4 and 5 years;
The incidence of reoperation due to dysfunction of prosthetic valve within 12 months and 2,3,4,5 years; | 12 months and within 2, 3, 4 and 5 years
  The incidence of reoperation due to dysfunction of prosthetic valve within 12 months and 2,3,4,5 years;
The incidence of readmission due to symptoms and signs of aortic valve disease within 12 months and 2,3,4,5 years; | 12 months and within 2, 3, 4 and 5 years
  The incidence of readmission due to symptoms and signs of aortic valve disease within 12 months and 2,3,4,5 years;
The incidence of prosthetic valve dysfunction at 12 months (moderate or severe stenosis or reflux by ultrasonography); | 12 months and within 2, 3, 4 and 5 years
  The incidence of prosthetic valve dysfunction at 12 months (moderate or severe stenosis or reflux by ultrasonography);
The incidence of thrombus in clinical and subclinical prosthetic heart valves at 12 months; | 12 months after aortic valve replacement
  The incidence of thrombus in clinical and subclinical prosthetic heart valves at 12 months;